CLINICAL TRIAL: NCT02452229
Title: Human Herpes Viruses in Burn Victims: A Systematic Review
Brief Title: Review of Human Herpes Viruses in Burns
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Other Study IDs: SHC-G-SR-HHV
Record Dates: First submitted 2015-05-14; First posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Human Herpes Virus; Herpes Simplex Virus; Varicella-zoster Virus; Chickenpox; Cytomegalovirus; Burns
MeSH Terms: conditions — Herpes Simplex; Chickenpox; Burns

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Burn patients: The included patient are burn victims who sustained a burn of at least 1 % total body surface are (TBSA); with no restriction on age.
  Interventions: Other: Review of the Literature for Human Herpes Virus infections

INTERVENTIONS:
Other: Review of the Literature for Human Herpes Virus infections — Review of the Medline database (PubMed and Ovid interface) for human herpes virus infections in burns as well as Web of Science interface.
  PRIMSA (preferred reporting items for systematic reviews and meta-analyses) guidelines and checklist were used.

SUMMARY:
Herpes simplex virus, cytomegalovirus and varicella zoster virus infection are purported to play a pivotal role in morbidity and mortality in burns. Thus far, there is no existing systematic review (Level of Evidence III or higher) describing the unique role as well as concurrent infections of these viruses in burns. The aim of this review is to point out the clinical differences between these human herpes virus subtypes, to outline established therapy approaches, and to provide evidence for virus related morbidity and mortality in burns.

DETAILED DESCRIPTION:
This systematic review was created according the PRIMSA (preferred reporting items for systematic reviews and meta-analyses) guidelines and checklist.

We performed an review of the medical literature to identify all studies that contain HSV, CMV and VZV infections in burns.Therefore, systematic review of the Medline database by using PubMed and Ovid interface was conducted. Also the Web of Science interface was used for systematic literature search.

On the PubMed interface, we used the following search terms: ("HSV"[All Fields] OR "herpes"[All Fields] OR "CMV"[All Fields] OR "cytomegalovirus"[All Fields] OR "VZV"[All Fields] OR "varicella-zoster"[All Fields]) AND ("burns"[MeSH Terms] OR "burns"[All Fields] OR "burn"[All Fields] OR "thermal trauma"[All Fields]). For Ovid we used: exp Burns/ AND (exp Herpes Zoster/ or exp Encephalitis, Herpes Simplex/ or exp Herpes Simplex/ or exp Herpes Simples Virus Vaccines/), exp Burns/ AND (exp Cytomegalovirus/ or exp Cytomegalovirus Infections/), exp Burns/ AND (exp Chickenpox/ or Herpesvirus 3. Human/ or exp Herpes Zoster/). And for Web of Science we used: (TS=(HSV OR herpes OR CMV OR cytomegalovirus OR VZV OR varicella-zoster) AND TS=(burn OR burns OR thermal trauma)) AND LANGUAGE: (English) AND DOCUMENT TYPES: (Article); Timespan: All years; Indexes: SCI-EXPANDED, SSCI, A&HCI, CPCI-S.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented with at least 1% TBSA burned
* Patients who presented with a viral infections during their hospitalization

Exclusion Criteria:

* Patients who had no burns
* Patients who had no viral infections during their hospitalization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every year, about 500,000 citizens of the United States of America were burned; 50,000 of them were admitted to Burn Center. Bacterial and viral infections including cellulitis, pneumonia, wound infections and septicemia are among the top ten complications of burn injuries. Severe burn injury causes an increased inflammatory response and an overall immunosuppression. As a result severely burned patients are more prone to infections and septicemia. Early treatment of sepsis and prevention of infections are key to reducing morbidity and improving the long-term outcome of burn victims.
Sampling Method: Non-Probability Sample
Enrollment: 10267 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of Human Herpes Virus (HHV) Infections | Participants will be followed for the duration of hospital stay, an expected average of 3 months.
  HHV include the herpes simplex virus type 1 (HSV-1), herpes simplex virus type 2 (HSV-2), varicella zoster virus (VZV), cytomegalovirus (CMV), Epstein-Barr viruses (EBV) and human herpes virus 6 to 8

SECONDARY OUTCOMES:
Treatment of Human Herpes Virus (HHV) Infections | Participants will be followed for the duration of hospital stay, an expected average of 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, FACS, Study Chair — Department of Surgery, University of Texas Medical Branch and Shriners Hospitals for Children, Galveston, Texas, USA

REFERENCES:
- [Background] Moher D, Liberati A, Tetzlaff J, Altman DG; PRISMA Group. Preferred reporting items for systematic reviews and meta-analyses: the PRISMA statement. Int J Surg. 2010;8(5):336-41. doi: 10.1016/j.ijsu.2010.02.007. Epub 2010 Feb 18. No abstract available. PMID 20171303